CLINICAL TRIAL: NCT01708044
Title: A Phase 1, Randomized, Placebo-Controlled Single-Blind, Dose-Ranging, 4-Way Crossover Study to Evaluate the Effect of Different Fixed Pramlintide: Insulin Dose Ratios on Postprandial Glycemic Control in Subjects With Type 1 Diabetes Mellitus
Brief Title: Effect of Different Fixed Pramlintide:Insulin Dose Ratios on Postprandial Glucose in T1DM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D5570C00001
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Type 1 Diabetes
Keywords: Pramlintide,; insulin,; type 1 diabetes,; reduction in postprandial glucose,; pramlintide:insulin dose-ratio
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — pramlintide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pramlintide 6 mcg per unit of insulin dose (Experimental): The pramlintide dose will be calculated based on the subjects' individual insulin units. Dose ratio to be examined is pramlintide 6 mcg for each unit of insulin.
  Interventions: Drug: Pramlintide acetate
- Pramlintide 9 mcg per unit of insulin dose (Experimental): The pramlintide dose will be calculated based on the subjects' individual insulin units. Dose ratio to be examined is pramlintide 9 mcg for each unit of insulin.
  Interventions: Drug: Pramlintide acetate
- Pramlintide 12 mcg per unit of insulin dose (Experimental): The pramlintide dose will be calculated based on the subjects' individual insulin units. Dose ratio to be examined is pramlintide 12 mcg for each unit of insulin.
  Interventions: Drug: Pramlintide acetate
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pramlintide acetate
  Arms: Pramlintide 12 mcg per unit of insulin dose; Pramlintide 6 mcg per unit of insulin dose; Pramlintide 9 mcg per unit of insulin dose
Other: Placebo — Placebo Comparator
  Arms: Placebo

SUMMARY:
To examine the effects of different fixed pramlintide:insulin dose ratios in subjects with type 1 diabetes on postprandial plasma glucose concentrations

ELIGIBILITY:
Inclusion Criteria:

* Is 18 to 70 years old
* Is male, or is female and meets all the following criteria:

  1. Not breastfeeding
  2. Negative pregnancy test result and, if of childbearing potential, must practice and be willing to continue to practice appropriate birth control
* Has been diagnosed with type 1 diabetes mellitus for at least 1 year and not achieving glycemic goal while on MDI of insulin
* Has HbA1c between 7.0% and 9.0%
* Has been on MDI of regular insulin, at a dose not to exceed 10 units/breakfast for at least 3 months or has been on continuous subcutaneous insulin infusion (CSII), at a dose not to exceed 10 units/breakfast, for at least 3 months and is willing to switch to an MDI insulin regimen for 1 day prior to enrollment and through the study
* Has a body mass index (BMI) <30 kg/m2

Exclusion Criteria:

* Has experienced recurrent severe hypoglycemia requiring assistance within 6 months before Visit 1 Screening
* Has a history of hypoglycemia unawareness
* Has a confirmed diagnosis of gastroparesis
* Has been treated, is currently being treated, or is expected to require or undergo treatment with the following medications:

  1. Any antihyperglycemic agent other than insulin
  2. Drugs that directly affect gastrointestinal motility (e.g., anticholinergic agents such as atropine)
  3. Drugs that slow the intestinal absorption of nutrients (e.g., α-glucosidase inhibitors.
* Has a clinically significant medical condition that could potentially affect study participation and/or personal well-being, as judged by the investigator, including but not limited to the following conditions:

  1. Hepatic disease
  2. Renal disease
  3. Gastrointestinal disease
  4. Pulmonary disease
  5. Organ transplantation
  6. Chronic infection (e.g., tuberculosis, human immunodeficiency virus, hepatitis B virus, or hepatitis C virus)
* Is currently treated or has been previously treated with SYMLIN/pramlintide or has participated in a SYMLIN/pramlintide clinical study within 3 months of Visit 1 (Screening).
* Has any clinically significant laboratory findings or medical history that may affect successful completion of the study and/or personal well-being
* Has donated blood within 2 months or is planning to donate blood during the study.
* Has had a major surgery or a blood transfusion within 2 months
* Has received any investigational drug within 1 month
* Has known allergies or hypersensitivity to any component of study treatment.
* Is an immediate family member of personnel directly affiliated with the study at the clinical study site, or is directly affiliated with the study at the clinical study site.
* Is employed by Amylin Pharmaceuticals, Inc (Amylin) (that is an employee, temporary contract worker, or designee responsible for the conduct of the study).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incremental area under the concentration-time curve (AUC(0-3 h)) of plasma glucose concentrations for each treatment | AUC 0-3 hrs compared to Placebo

SECONDARY OUTCOMES:
Incremental AUC (0-3 h) of plasma glucagon | 0-3 hrs compared to Placebo
Absolute AUC (0-3 h), peak plasma concentration (Cmax), Cave, and Tmax of glucagon of plasma glucose. | 0-3 hrs compared to Placebo
PK of pramlintide | 0-3 hrs compared to Placebo
Safety | 0-3 hrs compared to Placebo

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Portland, Oregon, United States

REFERENCES:
- [Derived] Riddle MC, Yuen KC, de Bruin TW, Herrmann K, Xu J, Ohman P, Kolterman OG. Fixed ratio dosing of pramlintide with regular insulin before a standard meal in patients with type 1 diabetes. Diabetes Obes Metab. 2015 Sep;17(9):904-7. doi: 10.1111/dom.12504. Epub 2015 Jul 8. PMID 26040429
- See also: ABA163_D5570C0001_CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2632&filename=ABA163_D5570C0001_CSR_Synopsis_Final_2014_08_27.pdf